CLINICAL TRIAL: NCT02686567
Title: The Use of the Transanal Drainage Tube for Prevention of Anastomotic Leakage After Laparoscopic Anterior Resection for Medium & Low Rectal Cancer
Brief Title: Use of the TDT for Prevention of Anastomotic Leakage After Laparoscopic Anterior Resection for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weidong Tong, Director of department of gastric and colorectal surgery, Daping Hospital, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDT20160214
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Anastomotic Leakage; Rectal Neoplasms
Keywords: transanal drainage tube; anastomotic leakage; laparoscopic anterior resection; rectal cancer
MeSH Terms: conditions — Anastomotic Leak; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with TDT (Active Comparator): with TDT
  Interventions: Procedure: with TDT
- without TDT (Active Comparator): without TDT
  Interventions: Procedure: without TDT

INTERVENTIONS:
Procedure: with TDT — After completion of the anastomosis and further DS construction if necessary, the surgeon would be notified to implement the intervention based on the randomizing results. In this group, a silicone tube (28Fr, Sumitomo Bakelite Co, Japan) was inserted through the anus and the tip of the tube was placed approximately 5 cm above the anastomosis at the end of the surgery in patients from the TDT group. The tube was fixed with a skin suture and connected to a drainage bag. TDT was planed to remove 3-7 days after surgery and early removal was allowed if the patient experienced intolerable pain.
  Other Names: with transanal drainage tube
  Arms: with TDT
Procedure: without TDT — After laparoscopic anterior resection and double-stapling technique anastomosis were finished, none additional proceduce was done.
  Other Names: without transanal drainage tube
  Arms: without TDT

SUMMARY:
The rate of anastomotic leakage after laparoscopic anterior resection（LAR） for medium & low rectal cancer is still high. the transanal drainage tube (TDT) was thought to be useful for deduce the rate. There were several studies, but most of them were not randomized controlled trial (RCT) studies. There was only one RCT study with enough samples, but it was designed for open anterior resection, and the patients underwent diverting stoma were excluded, so there was the selection bias. LAR now is thought to been with the same effect, and it is safe and feasible. So a RCT investigation for the use of TDT for prevention of anastomotic leakage after LAR for medium & low rectal cancer is needed.

DETAILED DESCRIPTION:
Patients were randomly assigned to two groups, the TDT and non-TDT group after the laparoscopic LAR and DST procedure was decided during operation. Randomization was obtained through a computer-generated random number sequence allocation. Surgeon blinding was performed to ensure all the intraoperative decisions made by the surgeon were not interfered with by the grouping. All the operative procedures fully complied with the guideline for the diagnosis and treatment of colorectal cancer and the technique of total mesorectal excision (TME). The preservation of the left colonic artery was judged by the surgeon according to his own experiences and assessment of the patient's conditions. When the anastomosis was accomplished, the discretion of DS construction was made by the surgeon based on assessing the risk factors of AL. Pelvic drainages were used in all cases in this study. After completion of the anastomosis and further DS construction if necessary, the surgeon would be notified to implement the intervention based on the randomizing results.

ELIGIBILITY:
Inclusion criteria: all consecutive 18 to 80 years old individuals diagnosed as primary rectal adenocarcinoma with the lower edge of the tumor less than 10 cm from the anal verge were considered eligible; with the classification of American Society of Anaesthesiologist (ASA) of I, II, or III; Laparoscopic LAR+ with double stapling technique (DST) was planned to perform for the patients. All the preoperative procedures should comply with the guideline for the diagnosis and treatment of colorectal cancer.

Exclusion criteria: The emergency operation for rectal cancer with obstruction, bleeding, or perforation would be excluded. Patients with inflammatory bowel disease (IBD), familial adenomatous polyposis (FAP), recurrent rectal cancer, or synchronous cancer would not be suitable. Patients with preoperative radiotherapy were excluded. Patients who underwent other types of surgeries for rectal cancer, including Hartmann's procedure, abdominoperineal resection (APR), intersphincteric resection ( ISR), et al. were excluded intraoperatively

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2016-02; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Incidence of AL | 30 days after surgery
  The primary endpoint was the AL within 30 days after surgery. AL is defined when the following symptoms were noticed: abdominal pain, fever, peritonitis, leukocytosis, procalcitonin (PCT) or c-reactive protein (CRP) increase, discharge of feces, pus, or gas from the drainage or vagina, septicemia with pelvic abscess. All clinically suspicious symptoms were confirmed by digital rectal examination, computed tomography (CT) scan or surgery when necessary. The severity grading of AL was defined according to the International Study Group of Rectal Cancer. In the present study, AL was referred to grade B and C, asymptomatic AL (grade A) was not considered because no active therapeutic intervention was required.

SECONDARY OUTCOMES:
Grades of AL | within 30 days after surgery
  The grades of AL, including grade B, grade C. The severity grading of AL is defined according to the International Study Group of Rectal Cancer
Postoperative Anal Pain Score | within 30 days after surgery
  Postoperative pain score. Numerical Rating Scale (NRS) for pains is used to assess the anal postoperative pain score of patients in the TDT group. NRS is the simplest and most commonly used scales for pain evaluation.The numerical scale is most commonly 0 to 10, with 0 being no pain and 10 being the worst pain imaginable. (for the details, please see the literature below FERREIRA-VALENTE M A, PAIS-RIBEIRO J L, JENSEN M P. Validity of four pain intensity rating scales[J]. Pain. 2011, 152(10): 2399-2404)
Incidence of TDT-related Adverse Events: bleeding | within 30 days after surgery
  TDT-related adverse events :bleeding

OTHER OUTCOMES:
Incidence of DT-related adverse events : iatrogenic colonic perforations | within 30 days after surgery
  DT-related adverse events : iatrogenic colonic perforations

CONTACTS AND LOCATIONS:
Overall Officials: Tong weidong, Professor, Principal Investigator — Daping Hospital, Third Military Medical University
Locations (1):
- Daping hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
after the paper published

REFERENCES:
- [Background] Xiao L, Zhang WB, Jiang PC, Bu XF, Yan Q, Li H, Zhang YJ, Yu F. Can transanal tube placement after anterior resection for rectal carcinoma reduce anastomotic leakage rate? A single-institution prospective randomized study. World J Surg. 2011 Jun;35(6):1367-77. doi: 10.1007/s00268-011-1053-3. PMID 21437746
- [Background] Matsuda M, Tsuruta M, Hasegawa H, Okabayashi K, Kondo T, Shimada T, Yahagi M, Yoshikawa Y, Kitagawa Y. Transanal drainage tube placement to prevent anastomotic leakage following colorectal cancer surgery with double stapling reconstruction. Surg Today. 2016 May;46(5):613-20. doi: 10.1007/s00595-015-1230-3. Epub 2015 Aug 1. PMID 26231480
- [Background] Shigeta K, Okabayashi K, Baba H, Hasegawa H, Tsuruta M, Yamafuji K, Kubochi K, Kitagawa Y. A meta-analysis of the use of a transanal drainage tube to prevent anastomotic leakage after anterior resection by double-stapling technique for rectal cancer. Surg Endosc. 2016 Feb;30(2):543-550. doi: 10.1007/s00464-015-4237-3. Epub 2015 Jun 20. PMID 26091985
- [Background] Ha GW, Kim HJ, Lee MR. Transanal tube placement for prevention of anastomotic leakage following low anterior resection for rectal cancer: a systematic review and meta-analysis. Ann Surg Treat Res. 2015 Dec;89(6):313-8. doi: 10.4174/astr.2015.89.6.313. Epub 2015 Nov 27. PMID 26665126
- [Background] Lee SY, Kim CH, Kim YJ, Kim HR. Impact of anal decompression on anastomotic leakage after low anterior resection for rectal cancer: a propensity score matching analysis. Langenbecks Arch Surg. 2015 Oct;400(7):791-6. doi: 10.1007/s00423-015-1336-5. Epub 2015 Aug 29. PMID 26318026
- [Background] Nishigori H, Ito M, Nishizawa Y, Nishizawa Y, Kobayashi A, Sugito M, Saito N. Effectiveness of a transanal tube for the prevention of anastomotic leakage after rectal cancer surgery. World J Surg. 2014 Jul;38(7):1843-51. doi: 10.1007/s00268-013-2428-4. PMID 24378550
- [Derived] Zhao S, Zhang L, Gao F, Wu M, Zheng J, Bai L, Li F, Liu B, Pan Z, Liu J, Du K, Zhou X, Li C, Zhang A, Pu Z, Li Y, Feng B, Tong W. Transanal Drainage Tube Use for Preventing Anastomotic Leakage After Laparoscopic Low Anterior Resection in Patients With Rectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2021 Dec 1;156(12):1151-1158. doi: 10.1001/jamasurg.2021.4568. PMID 34613330